CLINICAL TRIAL: NCT05016349
Title: Why Antiprogestrone (Mifepristone) and Cyp 26 Inhibitor Must be Combined With Tamoxifen or ( Tamoxifen and Retinoic Acid) for Treating Early Breast Cancer
Brief Title: Investigating the Potential Role of a Novel Quadrate Combination Therapy Mifepristone(Antiprogestrone), Tamoxifen, Retinoic Acid and Cannabidiol ( Selective Cyp 26 Inhibitor) for Treating Early Breast Cancer.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mahmoud Ramadan mohamed Elkazzaz (Other)
Collaborators: Ministry of Health, Saudi Arabia (Other Government)
Responsible Party: Sponsor-Investigator, Mahmoud Ramadan mohamed Elkazzaz, Clinical Researcher, Kafrelsheikh University
Organization: Kafrelsheikh University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: New theory(Tamoxifen&retinoic)
Record Dates: First submitted 2021-08-17; First posted 2021-08-23 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Breast Cancer Female
MeSH Terms: interventions — Tretinoin; Isotretinoin; Tocopherols; Mifepristone; Cannabidiol; Alitretinoin; Tamoxifen; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- All trans-retinoic acid, Mifepristone Cannabidiol (Epidiolex) and tamoxifen (Experimental): Patients will receive oral All trans-retinoic acid and Mifepristone daily for 2 weeks ,after which daily oral Cannabidiol (Epidiolex) is added to the regimen for 2 weeks , after which daily oral tamoxifen is added to the regimen. Patients continue treatment for up to 28 weeks, with tamoxifen continued after the study if medically appropriate.
  Interventions: Drug: All trans-retinoic acid; Drug: Mifepristone; Drug: Cannabidiol; Drug: Tamoxifen
- Mifepristone, Cannabidiol (Epidiolex) , All trans-retinoic acid and tamoxifen (Experimental): Patients will receive oral Mifepristone daily for 4 weeks ,after which daily oral All trans-retinoic acid, tamoxifen and Cannabidiol (Epidiolex) is added to the regimen , a. Patients continue treatment for up to 28 weeks, with tamoxifen continued after the study if medically appropriate.
  Interventions: Drug: All trans-retinoic acid; Drug: Mifepristone; Drug: Cannabidiol; Drug: Tamoxifen
- Mifepristone , All trans-retinoic acid, Cannabidiol (Epidiolex) and tamoxifen (Experimental): Patients will receive oral Mifepristone, All trans-retinoic acid and Cannabidiol (Epidiolex) daily for 4 weeks ,after which daily oral tamoxifen is added to the regimen , a. Patients continue treatment for up to 28 weeks, with tamoxifen continued after the study if medically appropriate.
  Interventions: Drug: All trans-retinoic acid; Drug: Mifepristone; Drug: Cannabidiol; Drug: Tamoxifen
- 9 cis retinoic acid, Mifepristone Cannabidiol (Epidiolex) and tamoxifen (Experimental): Patients will receive oral Mifepristone, 9 cis retinoic acid and Cannabidiol (Epidiolex) daily for 4 weeks ,after which daily oral tamoxifen is added to the regimen , a. Patients continue treatment for up to 28 weeks, with tamoxifen continued after the study if medically appropriate.
  Interventions: Drug: Mifepristone; Drug: Cannabidiol; Drug: 9 cis retinoic acid; Drug: Tamoxifen
- Mifepristone, 13 cis retinoic acid , Cannabidiol (Epidiolex) and tamoxifen (Experimental): Patients will receive oral Mifepristone, 13 cis retinoic acid and Cannabidiol (Epidiolex) daily for 4 weeks ,after which daily oral tamoxifen is added to the regimen , a. Patients continue treatment for up to 28 weeks, with tamoxifen continued after the study if medically appropriate.
  Interventions: Drug: 13-Cis Retinoic Acid plus Tocopherol; Drug: Mifepristone; Drug: Cannabidiol; Drug: Tamoxifen
- 9 cis retinoic acid , Mifepristone Cannabidiol (Epidiolex) and tamoxifen (Experimental): Patients will receive oral 9 cis retinoic acid and Mifepristone daily for 2 weeks ,after which daily oral Cannabidiol (Epidiolex) is added to the regimen for 2 weeks , after which daily oral tamoxifen is added to the regimen. Patients continue treatment for up to 28 weeks, with tamoxifen continued after the study if medically appropriate.
  Interventions: Drug: Mifepristone; Drug: Cannabidiol; Drug: 9 cis retinoic acid; Drug: Tamoxifen
- 13 cis retinoic acid , Mifepristone Cannabidiol (Epidiolex) and tamoxifen (Experimental): Patients will receive oral Mifepristone, 13 cis retinoic acid and Cannabidiol (Epidiolex) daily for 4 weeks ,after which daily oral tamoxifen is added to the regimen , a. Patients continue treatment for up to 28 weeks, with tamoxifen continued after the study if medically appropriate.
  Interventions: Drug: 13-Cis Retinoic Acid plus Tocopherol; Drug: Mifepristone; Drug: Cannabidiol; Drug: Tamoxifen
- Standard therapy (Sham Comparator): Patients will receive the approved standard therapy
  Interventions: Drug: Standard therapy

INTERVENTIONS:
Drug: All trans-retinoic acid — Vesanoid will be supplied orally at the total dosage of 45mg/m2/d (two daily administrations of 22.5 mg/m2 each). Treatment will last 28 days
  Other Names: Vesanoid
  Arms: All trans-retinoic acid, Mifepristone Cannabidiol (Epidiolex) and tamoxifen; Mifepristone , All trans-retinoic acid, Cannabidiol (Epidiolex) and tamoxifen; Mifepristone, Cannabidiol (Epidiolex) , All trans-retinoic acid and tamoxifen
Drug: 13-Cis Retinoic Acid plus Tocopherol — 13-Cis Retinoic Acid (50 mg/m2/d) Tocopherol (800 mg/day) supplied orally at the total dosage of 50 mg/m2/d (two daily administrations of 25 mg/m2 each). Treatment will last 28 days
  Arms: 13 cis retinoic acid , Mifepristone Cannabidiol (Epidiolex) and tamoxifen; Mifepristone, 13 cis retinoic acid , Cannabidiol (Epidiolex) and tamoxifen
Drug: Mifepristone — Mifepristone 200mg capsules daily for 28 days
  Arms: 13 cis retinoic acid , Mifepristone Cannabidiol (Epidiolex) and tamoxifen; 9 cis retinoic acid , Mifepristone Cannabidiol (Epidiolex) and tamoxifen; 9 cis retinoic acid, Mifepristone Cannabidiol (Epidiolex) and tamoxifen; All trans-retinoic acid, Mifepristone Cannabidiol (Epidiolex) and tamoxifen; Mifepristone , All trans-retinoic acid, Cannabidiol (Epidiolex) and tamoxifen; Mifepristone, 13 cis retinoic acid , Cannabidiol (Epidiolex) and tamoxifen; Mifepristone, Cannabidiol (Epidiolex) , All trans-retinoic acid and tamoxifen
Drug: Cannabidiol — Liquid taken orally for daily for 28 days
  Other Names: Epidiolex
  Arms: 13 cis retinoic acid , Mifepristone Cannabidiol (Epidiolex) and tamoxifen; 9 cis retinoic acid , Mifepristone Cannabidiol (Epidiolex) and tamoxifen; 9 cis retinoic acid, Mifepristone Cannabidiol (Epidiolex) and tamoxifen; All trans-retinoic acid, Mifepristone Cannabidiol (Epidiolex) and tamoxifen; Mifepristone , All trans-retinoic acid, Cannabidiol (Epidiolex) and tamoxifen; Mifepristone, 13 cis retinoic acid , Cannabidiol (Epidiolex) and tamoxifen; Mifepristone, Cannabidiol (Epidiolex) , All trans-retinoic acid and tamoxifen
Drug: 9 cis retinoic acid — 9 cis retinoic acid will be supplied orally at the total dosage of 45mg/m2/d (two daily administrations of 22.5 mg/m2 each). Treatment will last 28 days
  Arms: 9 cis retinoic acid , Mifepristone Cannabidiol (Epidiolex) and tamoxifen; 9 cis retinoic acid, Mifepristone Cannabidiol (Epidiolex) and tamoxifen
Drug: Tamoxifen — Patients will be given 10mg Tamoxifen twice a day. Treatment will last 28 days
  Arms: 13 cis retinoic acid , Mifepristone Cannabidiol (Epidiolex) and tamoxifen; 9 cis retinoic acid , Mifepristone Cannabidiol (Epidiolex) and tamoxifen; 9 cis retinoic acid, Mifepristone Cannabidiol (Epidiolex) and tamoxifen; All trans-retinoic acid, Mifepristone Cannabidiol (Epidiolex) and tamoxifen; Mifepristone , All trans-retinoic acid, Cannabidiol (Epidiolex) and tamoxifen; Mifepristone, 13 cis retinoic acid , Cannabidiol (Epidiolex) and tamoxifen; Mifepristone, Cannabidiol (Epidiolex) , All trans-retinoic acid and tamoxifen
Drug: Standard therapy — Patients will receive the approved standard therapy tamoxifen
  Arms: Standard therapy

SUMMARY:
Investigating the potential role of a novel quadrate combination therapy Mifepristone(Antiprogestrone), Tamoxifen, Retinoic acid and Cannabidiol ( selective cyp 26 inhibitor) for treating early breast cancer.

Breast cancer is the main cause of mortality among women. The disease presents high recurrence mainly due to incomplete efficacy of primary treatment in killing all cancer cells. Therapy resistance remains a major problem in estrogen receptor-α (ERα)-positive breast cancer. Half of estrogen receptor-positive breast cancers contain a subpopulation of cytokeratin 5 (CK5)-expressing cells that are therapy resistant and exhibit increased cancer stem cell (CSC) properties. Here, we propose a testable hypothesis that treatment of breast cancer with tamoxifen or retinoic acid or a combination of the two, may result in induction or conversion of some ER-positive breast cancer cells to ER-negative cancer cells expressing the basal cytokeratin-5 (CK5) via stimulation of progesterone receptors effect, and production . Therefore, we raised an issue with the answer " Why Antiprogestrone such Mifepristone and cyp 26 inhibitors must be combined with Tamoxifen or its combination with retinoic acid in the era of oncology for treating early breast cancer" .In fact, limited evidence has indicated that induction of CK5+ cells in ERα+ breast cancer is a unique effect of progestin (Prg) but many studies have demonstrated that progesterone (P4) increases CK5+ breast cancer cells. In case-cohort study of 405 incident breast cancer cases, elevated circulating progesterone levels were associated with a 16% increase in the risk of breast cancer. A study demonstrated that tamoxifen induced progesterone receptors (PGR) in short term treatment. Another study showed that High progesterone receptor expression correlates to the effect of adjuvant tamoxifen in premenopausal breast cancer patients. These CK5-positive cells are therapy resistant and have increased tumor-initiating potential. Also, previous work has shown that retinoic acid, a chemical that results from the body's natural breakdown of vitamin A, should act against these CK5+ cells, but clinical trials of retinoids against breast cancer have been largely unsuccessful .Therefore we suggest that combination of retinoiac acid and tamoxifen was unsucssecful in treating breast cancer owing its ability to induce progesterone receptors and production leading to increasing numbers of CK5-positive cells which are therapy resistant . Although retinoid fenretinide reduced the accumulation of CK5+ cells during estrogen depletion. A study investigated the effects of all-trans-RA (atRA) on progesterone production in immature rat GCs cultured without gonadotropin. demonstrated that atRA enhanced progesterone production by upregulating the levels of steroidogenic acute regulatory protein (StAR) and cytochrome P450scc (Cyp11a1). Here, we suggest that tamoxifen or its combination with retinoic acid must be combined with anti-progesterone (Mifepristone) to achieve treatment with significant effect against early breast cancer. Moreover, Numerous studies have shown that CYP2D6 variant carriers (around 50% CYP2D6 variant carriers in Chinese population) will not benefit a lot from tamoxifen, and combined use of CYP2D6 inhibitors will further affect the efficacy of tamoxifen. In addition, All-trans-retinoic acid acts as an inducer of CYP26A1 expression. Which is the second expected cause of unsuccessful trial of Tamoxifen and retinoic acid in breast cancer treatment. Furthermore, The CYP26 inhibitor also induced expression of atRA-responsive genes. All-trans retinoic acid (ATRA) significantly inhibited aromatase activity in a concentration-dependent manner in microsomes isolated from JEG-3 human placental carcinoma cells. One study found that high retinol was significantly. associated with reduced breast cancer risk. Another found a significant trend of reduced retinol levels with more advanced disease stage. A study showed that intake of vitamin A and retinol could reduce breast cancer risk. Therefore we will take the benefit of cyp 26 inhibitor in this trial by combining Cannabidiol, a major phytocannabinoid, as a potent atypical inhibitor for CYP2D6.

DETAILED DESCRIPTION:
The study is a randomized interventional comparative Phase II trial. which will Investigating and test the safety and effectiveness of a Novel Quadrate Combination Therapy Mifepristone(Antiprogestrone), Tamoxifen, Retinoic Acid and Cannabidiol ( Selective Cyp 26 Inhibitor) to learn whether this novel combination therapy works in treating Treating Early Breast Cancer. The primary objective of the study is to; 1) evaluate the anti-tumor activity of this combination therapy within the context of a phase II study Other objectives are: 2) to determine the effect of this novel combination therapy on cytokeratin 5 (CK5)-expressing cells;3) and to determine the expression of CK5 biomarkers of breast carcinogenesis before and after treatment.160 adult female patients with breast cancer and fulfilling the below outlined inclusion criteria will be enrolled into the study.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent/assent for the trial.
2. Be 18 years of age on day of signing informed consent
3. Confirmed diagnosis of breast cancer positive at least for CEA tumor marker at above normal threshold level.
4. e willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion. Newly-obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on Day 1. Subjects for whom newly-obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived specimen only upon agreement from the Sponsor.
5. Demonstrate adequate organ function as defined in Table 1, all screening labs should be performed within 10 days of treatment initiation.

   Table 1 Adequate Organ Function Laboratory Values System Laboratory Value Hematological Absolute neutrophil count (ANC) ≥1,500 /mcL Platelets ≥100,000 / mcL Hemoglobin ≥9 g/dL or ≥5.6 mmol/L without transfusion or EPO dependency (within 7 days of assessment) Renal Serum creatinine OR Measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤1.5 X upper limit of normal (ULN) OR

   ≥60 mL/min for subject with creatinine levels > 1.5 X institutional ULN Hepatic Serum total bilirubin ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN OR

   ≤ 5 X ULN for subjects with liver metastases Albumin >2.5 mg/dL Coagulation International Normalized Ratio (INR) or Prothrombin Time (PT)

   Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants

   ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants a Creatinine clearance should be calculated per institutional standard.

   Exclusion Criteria:
   * Pregnant
   * Treatment including radiation therapy, chemotherapy, biotherapy and/or hormonal therapy for the currently diagnosed breast cancer prior to study entry.
   * Any medical or other condition that in the Investigator's opinion renders the patient unsuitable for this study due to unacceptable risk
   * Psychiatric disorders or altered mental status precluding understanding of the informed consent process and/or completion of the necessary studies
   * Gastrointestinal disorders that may interfere with absorption of the study drug.
   * Co-existing active infection or serious concurrent illness
   * Current uncontrolled illness, for instance sepsis, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia
   * Current use of antiretroviral therapy
   * Participants with psychiatric illness or social situations that would limit compliance with study requirements
   * Current hepatocellular carcinoma, liver metastases, or documented history of difficult to control diabetes

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Cytokeratin 5 (CK5)-expression | Baseline to 4 weeks
  Cytokeratin 5 (CK5)-expression
To evaluate and compare the pathological complete response (pCR) rates | Up to 1 month after treatment

SECONDARY OUTCOMES:
To evaluate the overall clinical response rate | Up to 1 month after treatment
Estradiol and progesterone levels in breast tissue and plasma assessed by liquid chromatography/tandem mass spectrometry | Up to 1 month after treatment
  Analysis will be pilot in nature and will provide descriptive statistics for each group or subgroup of subjects, supplying results which may be used to plan future studies.
Retinoic acid, TAM and their metabolites levels in breast tissue and plasma | Up to 1 month after treatment
  Analysis will be pilot in nature and will provide descriptive statistics for each group or subgroup of subjects, supplying results which may be used to plan future studies.
Effect on level of serum tumor markers compared to baseline | Weekly for 4 weeks
  Commonly measured tumor markers associated with breast cancer, primarily CA 15-3, CA 27.29, and CEA, at baseline and at study termination

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Elkazzaz, Principal Investigator — New Damietta University Hospital; Amr Ahmed, Principal Investigator — Ministry of Health